CLINICAL TRIAL: NCT05427916
Title: Prospective Randomized Evaluation of the Effect of Avance® Solo Negative Pressure Wound Therapy System or Optifoam® Gentle Post-Op Dressing on "High Risk" Closed Surgical Incisions; Freedom From Wound Complication Study
Brief Title: Closed Incision Negative Pressure Wound Therapy vs. Foam as Post Operative Dressing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Site decided not to continue
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, John Lantis, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-22-00329
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Diabetes; Morbid Obesity; Lymphedema; Orthopedic Disorder
MeSH Terms: conditions — Diabetes Mellitus; Obesity, Morbid; Lymphedema; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Negative Pressure Wound Therapy (Experimental): Negative pressure to the incision site and managing exudate generated by the incision.
  Interventions: Device: Avance Solo
- Optifoam (Active Comparator): This foam is standard of care and is currently stocked by the operating rooms at Mount Sinai hospital and indicated for use in high risk wounds
  Interventions: Other: Optifoam

INTERVENTIONS:
Device: Avance Solo — Avance® Solo will include the collective description for a complete device capable of delivering negative pressure to the incision site and managing exudate generated by the incision.
  Arms: Negative Pressure Wound Therapy
Other: Optifoam — Optifoam is a silicone backed foam that is conformable, with a border that is waterproof, flexible and breathable for increased comfort, with a wear time of up to seven days. It is a standard of care product that is given to patients for surgical wounds.
  Arms: Optifoam

SUMMARY:
The primary objective is to assess the frequency of a wound healing complication, in a closed incisional wound in a "high risk" surgical incision when treated with Negative Pressure Wound Therapy versus a highly absorbent antimicrobial post - operative absorbent dressing.

DETAILED DESCRIPTION:
A healing complication is defined as presence of at least one of the following conditions: infection (superficial or deep), dehiscence (partial, superficial, or deep), or delayed healing (incision not 100% closed within 7 days of the first surgical procedure), drainage form the wound after 96 hours post operatively.

The secondary objectives are to assess any changes in the following assessments of the surgical incision weekly over the treatment period:

* Surrounding skin condition
* Incision complications, infection or clinical signs of infection
* to assess the number and type of these complications individually including other postsurgical complications: skin necrosis, cellulitis, abscess, suture abscess, seroma, periwound edema or hematoma occurring within 21, 42, and 90 days postoperatively
* Pain during dressing changes

Assessment of the following at dressing changes:

* Duration/wear time
* Ease of use; difficulty with sleep
* Damage to surrounding skin on removal
* Assessment of re-epithelialization/closure
* Patient comfort during wear; ease of ambulation
* Conformability of dressing
* Exudate management
* Reasons for removal

To assess the overall comparison of Avance® Solo to the standard of care foam dressing.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years of age.
* Males and females - provided they are not pregnant and if of reproductive age are using contraception.
* Have a closed surgical incision post-surgery/closure (<24 hours after).
* The patient is able to understand the evaluation and is willing to consent to the evaluation.
* Undergoing appropriate: wound "high risk" surgery.
* Foot and ankle surgery.
* Vascular groin incision.
* Long leg vein harvest incision.
* Closed forefoot and major amputation surgery.
* Possibly: breast augmentation and reduction surgery.
* HIV and hepatitis positive patients will not be excluded from this study.
* Renal failure patients will not be excluded.
* Patient on metabolic agent, immunosuppressants, or steroid therapy will not be excluded from this study.

Exclusion Criteria:

* Incisions in excess of effective dressing pad size provided.
* Patients with a known history of poor compliance with medical treatment.
* Patients who have participated in this trial previously and who were withdrawn.
* Patients with known allergies to product components (silicone adhesives and polyurethane films (direct contact with incision), acrylic adhesives (direct contact with skin), polyethylene fabrics and super-absorbent powders (polyacrylates) (within the dressing).
* Incisions where daily inspection is required underneath the dressing.
* Incisions which have an infection which is not being treated with systemic antibiotics.
* Incisions which are actively bleeding.
* Exposure of blood vessels, organs, bone or tendon at the base of the reference incision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Lantis, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Lauren Rodio, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data. Any purpose. Proposals should be directed to john.lantis@mountsinai.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 6/1/22, with first enrollment on 7/12/22. Recruitment continued until study was terminated on 5/1/23.
Period: Overall Study
Arm/Group | Negative Pressure Wound Therapy | Optifoam
Started | 12 | 8
Completed | 0 | 0
Not Completed | 12 | 8
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 6 | 0
Not completed — Active arm terminated; trial was ended. | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Pressure Wound Therapy | Optifoam | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Continuous [Median (Full Range); unit: years] | 58 [45 to 82] | 71 [51 to 83] | 64 [45 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 2 | 3 | 5
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Healing Complication
Description: Healing complications are defined as the presence of at least one of the following conditions: infection (superficial or deep), dehiscence (partial, superficial, or deep), or delayed healing (incision not 100% closed within 7 days of the first surgical procedure)
Time Frame: 21 days
Population: Data not collected. Study terminated before endpoint data collection.
Arm/Group | Negative Pressure Wound Therapy | Optifoam
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Skin Necrosis Complications
Description: Incisional complication as assessed by number of skin necrosis complications
Time Frame: 90 days
Population: Data not collected. Study terminated before endpoint data collection.
Arm/Group | Negative Pressure Wound Therapy | Optifoam
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Cellulitis Complications
Description: Incisional complication as assessed by number of cellulitis complications
Time Frame: 90 days
Population: Data not collected. Study terminated before endpoint data collection.
Arm/Group | Negative Pressure Wound Therapy | Optifoam
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Abscess Complications
Description: Incisional complication as assessed by number of abscess complications
Time Frame: 90 days
Population: Data not collected. Study terminated before endpoint data collection.
Arm/Group | Negative Pressure Wound Therapy | Optifoam
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Suture Abscess Complications
Description: Incisional complication as assessed by number of suture abscess complications
Time Frame: 90 days
Population: Data not collected. Study terminated before endpoint data collection.
Arm/Group | Negative Pressure Wound Therapy | Optifoam
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Seroma Complications
Description: Incisional complication as assessed by number of seroma complications
Time Frame: 90 days
Population: Data not collected. Study terminated before endpoint data collection.
Arm/Group | Negative Pressure Wound Therapy | Optifoam
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Periwound Edema Complications
Description: Incisional complication as assessed by number of periwound edema complications
Time Frame: 90 days
Population: Data not collected. Study terminated before endpoint data collection.
Arm/Group | Negative Pressure Wound Therapy | Optifoam
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Hematoma Complications
Description: Incisional complication as assessed by number of hematoma complications
Time Frame: 90 days
Population: Data not collected. Study terminated before endpoint data collection.
Arm/Group | Negative Pressure Wound Therapy | Optifoam
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Pain During Dressing Changes
Description: Patient reported as none, mild, moderate, or severe
Time Frame: 90 days
Population: Data not collected. Study terminated before endpoint data collection.
Arm/Group | Negative Pressure Wound Therapy | Optifoam
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Patient Satisfaction
Description: Patient Satisfaction Question that the patient will rank on a min/max scale of 0 to 7, higher score indicates higher satisfaction
Time Frame: 90 days
Population: Data not collected. Study terminated before endpoint data collection.
Arm/Group | Negative Pressure Wound Therapy | Optifoam
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Two weeks.
Arm/Group | Negative Pressure Wound Therapy | Optifoam
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 3/12 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Negative Pressure Wound Therapy (N=12) | Optifoam (N=8)
Excessive serosanguinoius fluid secretion (Blood and lymphatic system disorders) | 1 | 0
Excessive bleeding (Blood and lymphatic system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT05427916/Prot_SAP_000.pdf